CLINICAL TRIAL: NCT02901795
Title: Fetal Heart Rate Variability Analysis for the Early Detection of Chorioamnionitis During Preterm Premature Rupture of Membranes
Brief Title: Early Detection of Chorioamnionitis in Preterm Premature Rupture of Membranes
Acronym: AiRPM
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC14_9772
Record Dates: First submitted 2016-09-05; First posted 2016-09-15 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Fetal Membranes, Premature Rupture
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
All included patients will have their fetal heart rate recording performed with an EDAN F3 fetal monitor that allowed the back up recording of the fetal heart rate beat to beat detection. Fetal heart rate variability analysis will be performed using Matalb® software.

DETAILED DESCRIPTION:
Preterm Premature Rupture Of Membranes (pPROM) complicates 2-3% of all pregnancies and is responsible for one-third of preterm birth. Since the membranes generally form a barrier to ascending infection, the second major complication (10-36%) of pPROM is the development of intrauterine infection, called chorioamnionitis. It involves infection/inflammation of the fetus and increases neonatal morbidity and mortality. Indeed, histological chorioamnionitis (microscopic evidence of polynuclear neutrophils on examination of the placenta), regardless the prematurity, creates an inflammatory fetal syndrome which is responsible for an increase rate of cerebral palsy, intracranial hemorrhage, sepsis, pneumonia, respiratory distress syndrome and necrotizing enterocolitis at birth.

During hospitalization, management of women who develop pPROM requires an individual assessment of the benefits and risks of continuing pregnancy versus immediate delivery to avoid chorioamnionitis. Numerous studies in recent years have failed to identify a satisfactory prenatal marker of infection to predict chorioamnionitis. It is now clearly recognized that new markers are needed to improve prediction of infection in cases of pPROM.

A retrospective study (under submission) based on 23 pregnant women with pPROM was performed in the University Hospital of Rennes between 2007 and 2012. For all the patients included, a computerized analysis of the fetal heart rate (Sonicaïd FetalCare Oxford 8002®) has been performed daily during the last six days before delivery and the last recording was made less than 24 hours before the delivery. This study found significant differences of fetal heart rate patterns from pPROM complicated by histological chorioamnionitis compared with pPROM without histological chorioamnionitis. Short term variation (p=0,003) and high variation episodes (p<0,001) decreased significantly in pPROM complicated by histological chorioamnionitis. An index based on the high variations episodes was performed and seems a promising tool for the early detection of chorioamnionitis during pPROM (sensitivity 90%, specificity 84.6%, positive predictive value 71.5%, negative predictive value 95.2%, AUC = 0.88, IC 95% 0.73 to 100).

These data are consistent with those observed in neonatology for the assessment of early-onset sepsis and the underlying pathophysiological mechanisms (decreased fetal heart rate variability and adaptability in response to the placental infection/inflammation). Therefore, fetal heart rate (FHR) characteristics could be a potential way of research still unexploited for the early detection of chorioamnionitis in cases of pPROM.

ELIGIBILITY:
Inclusion Criteria:

* pPROM between 26 to 34 WG clinically proven or confirmed by a positive IGBP-1 protein test in a vaginal sample
* 18 years old or older
* singleton pregnancy

Exclusion Criteria:

* multiple pregnancy
* intra-uterine growth restriction defined by a fetal weight under the 10th percentile (AUDIPOG)
* active smoking
* gestational diabetes or pre-existing diabetes mellitus
* maternal pathology :

  * congenital or acquired heart defect
  * pulmonary embolism in progress or under treatment
  * pulmonary hypertension
  * renal insufficiency
  * Chronic obstructive pulmonary disease
  * systemic lupus erythematosus, multiple sclerosis, Sjögren's syndrome
* heart, neurological or genetic fetal proven malformations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women with pPROM between 26 to 34 WG clinically proven or confirmed by a positive IGBP-1 protein test in a vaginal sample
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-21 (Actual)

PRIMARY OUTCOMES:
The performance indicator | up to delivery
  area under ROC curve of the high variation index for the early diagnosis of histologically proven chorioamnionitis during pPROM.
The performance indicator | up to delivery
  sensibility, specificity of the high variation index for the early diagnosis of histologically proven chorioamnionitis during pPROM.
The performance indicator | up to delivery
  positive predictive value of the high variation index for the early diagnosis of histologically proven chorioamnionitis during pPROM.
The performance indicator | up to delivery
  negative predictive value of the high variation index for the early diagnosis of

CONTACTS AND LOCATIONS:
Overall Officials: Linda Lassel, MD, Principal Investigator — CHU Rennes Hopital Sud
Locations (4):
- France (4):
  - CHU Rennes Hôpital Sud, Rennes, Brittany Region
  - Service de Gynecologie obstétrique, Angers
  - Service de gynecologique-obstétrique, Nantes
  - Service de Gynecologie Obstétrique, Poitiers